CLINICAL TRIAL: NCT00714285
Title: Immunogenicity and Safety Study of a GSK Influenza Vaccine Candidate GSK 2115160A in Adults.
Brief Title: Immunogenicity and Safety Study of a GSK Influenza Vaccine Candidate in Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 111295
Record Dates: First submitted 2008-07-11; First posted 2008-07-14 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2017-03

CONDITIONS: Influenza
Keywords: Primary study; immunogenicity; safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Quadrivalent influenza vaccine GSK 2115160A Group 1 (Experimental): Subjects in this group received 1 full dose of GSK Biologicals' quadrivalent influenza vaccine, administered intramuscularly in the deltoid region of the non-dominant arm, at Day 0
  Interventions: Biological: GSK Biologicals' quadrivalent influenza vaccine
- Quadrivalent influenza vaccine GSK 2115160A Group 2 (Experimental): Subjects in this group received 1 low dose of GSK Biologicals' quadrivalent influenza vaccine, administered intramuscularly in the deltoid region of the non-dominant arm, at Day 0
  Interventions: Biological: GSK Biologicals' quadrivalent influenza vaccine
- Trivalent influenza vaccine GSK 2115160A Group 1 (Active Comparator): Subjects in this group received 1 low dose of GSK Biologicals' trivalent influenza vaccine, administered intramuscularly in the deltoid region of the non-dominant arm, at Day 0
  Interventions: Biological: GSK Biologicals' trivalent influenza vaccine
- Trivalent influenza vaccine GSK 2115160A Group 2 (Active Comparator): Subjects in this group received 1 full dose of GSK Biologicals' trivalent influenza vaccine, administered intramuscularly in the deltoid region of the non-dominant arm, at Day 0
  Interventions: Biological: GSK Biologicals' trivalent influenza vaccine

INTERVENTIONS:
Biological: GSK Biologicals' quadrivalent influenza vaccine — Single intramuscular dose on Day 0.
  Arms: Quadrivalent influenza vaccine GSK 2115160A Group 1; Quadrivalent influenza vaccine GSK 2115160A Group 2
Biological: GSK Biologicals' trivalent influenza vaccine — Single intramuscular dose on Day 0.
  Arms: Trivalent influenza vaccine GSK 2115160A Group 1; Trivalent influenza vaccine GSK 2115160A Group 2

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of GSK influenza vaccine candidate compared to a licensed trivalent influenza vaccine in adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 18 and 60 years of age at the time of the vaccination.
* Written informed consent obtained from the subject.
* If the subject is female, she must be of non-childbearing potential, if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 3 months prior to administration of the vaccine.
* Administration of a vaccine not foreseen in the study protocol from 30 days before vaccination up to 21 days post vaccination.
* Confirmed influenza infection within a year preceding the study start.
* Administration of an influenza vaccine during Northern Hemisphere season 2007-2008.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* History of hypersensitivity to a previous dose of influenza vaccine
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* History of administration of experimental/licensed vaccine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2008-07-14; Primary Completion 2009-01-28 (Actual); Study Completion 2009-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Beran J, Peeters M, Dewe W, Raupachova J, Hobzova L, Devaster JM. Immunogenicity and safety of quadrivalent versus trivalent inactivated influenza vaccine: a randomized, controlled trial in adults. BMC Infect Dis. 2013 May 20;13:224. doi: 10.1186/1471-2334-13-224. PMID 23688546
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 111295 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111295 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111295 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111295 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111295 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111295 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111295 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Started | 105 | 105 | 105 | 105
Completed | 105 (Completed upto Day 180) | 102 (Completed upto Day 180) | 105 (Completed upto Day 180) | 104 (Completed upto Day 180)
Not Completed | 0 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 1
Not completed — Migrated/moved from study area | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2 | Total
Number analyzed (Participants) | 105 | 105 | 105 | 105 | 420
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (11.85) | 37.6 (12.30) | 36.6 (12.87) | 37.4 (12.51) | 37.5 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 66 | 66 | 58 | 251
  Male | 44 | 39 | 39 | 47 | 169

OUTCOME MEASURES:

1. Primary Outcome: Serum Haemagglutination-inhibition (HI) Antibody Titers, Against Each of the Vaccine Influenza Virus Strains.
Description: Antibody titers were expressed as Geometric mean titers (GMTs).The vaccine influenza strains included A/Solomon Islands,A/Wisconsin,B/Malaysia and B/Jiangsu antigens.
Time Frame: At Day 0 and Day 21
Population: Analysis was performed on According To Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 104 | 104 | 104 | 105
Titer
  A/Solomon Islands strain, Day 0 | 21.4 [16.1 to 28.4] | 22.2 [16.6 to 29.5] | 23.3 [17.5 to 31.0] | 18.4 [14.3 to 23.7]
  A/Solomon Islands strain, Day 21 | 130.0 [106.1 to 159.4] | 150.6 [118.4 to 191.5] | 160.4 [129.1 to 199.3] | 133.8 [105.6 to 169.7]
  A/Wisconsin strain, Day 0 | 29.3 [23.0 to 37.3] | 25.7 [19.8 to 33.3] | 30.7 [23.7 to 39.8] | 29.0 [22.5 to 37.4]
  A/Wisconsin strain, Day 21 | 162.1 [138.0 to 190.4] | 189.5 [158.9 to 226.0] | 197.9 [169.1 to 231.7] | 156.3 [127.5 to 191.6]
  B/Malaysia strain, Day 0 | 32.2 [24.8 to 41.8] | 26.6 [20.2 to 35.0] | 23.2 [17.7 to 30.4] | 27.2 [20.6 to 35.8]
  B/Malaysia strain, Day 21 | 192.8 [159.6 to 232.9] | 213.0 [174.0 to 260.9] | 187.0 [151.9 to 230.3] | 188.5 [150.0 to 237.0]
  B/Jiangsu strain, Day 0 | 19.6 [15.6 to 24.8] | 19.5 [15.4 to 24.5] | 23.4 [18.3 to 29.7] | 19.2 [15.2 to 24.3]
  B/Jiangsu strain, Day 21 | 179.1 [151.4 to 211.9] | 158.3 [130.7 to 191.9] | 59.2 [47.3 to 74.0] | 43.4 [34.5 to 54.6]

2. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against the Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40 or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer. The vaccine influenza strains included A/Solomon Islands, A/Wisconsin, B/Malaysia and B/Jiangsu antigens.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 104 | 104 | 104 | 105
Subjects
  A/Solomon Islands strain | 59 | 60 | 57 | 63
  A/Wisconsin strain | 63 | 69 | 67 | 62
  B/Malaysia strain | 60 | 68 | 59 | 62
  B/Jiangsu strain | 79 | 82 | 28 | 20

3. Secondary Outcome: HI Antibody Seroconversion Factors Against the Vaccine Influenza Strains
Description: Seroconversion factors were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The Influenza vaccine strains included A/Solomon Islands, A/Wisconsin, B/Malaysia and B/Jiangsu antigens.
Time Frame: Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 104 | 104 | 104 | 105
Fold increase
  FA/Solomon Islands strain | 6.1 [4.6 to 8.0] | 6.8 [5.0 to 9.2] | 6.9 [5.0 to 9.4] | 7.3 [5.3 to 9.9]
  A/Wisconsin strain | 5.5 [4.4 to 6.9] | 7.4 [5.8 to 9.4] | 6.4 [5.0 to 8.3] | 5.4 [4.1 to 7.0]
  B/Malaysia strain | 6.0 [4.7 to 7.7] | 8.0 [6.1 to 10.5] | 8.1 [5.9 to 11.0] | 6.9 [5.2 to 9.3]
  B/Jiangsu strain | 9.1 [7.2 to 11.5] | 8.1 [6.6 to 10.0] | 2.5 [2.1 to 3.0] | 2.3 [1.9 to 2.6]

4. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against the Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a subject with a serum HI titer ≥1:40 that usually is accepted as indicating protection. The Influenza vaccine strains included A/Solomon Islands, A/Wisconsin, B/Malaysia and B/Jiangsu antigens.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 104 | 104 | 104 | 105
Subjects
  A/Solomon Islands strain, Day 0 | 39 | 44 | 42 | 37
  A/Solomon Islands strain, Day 21 | 96 | 92 | 97 | 95
  A/Wisconsin strain, Day 0 | 53 | 48 | 56 | 58
  A/Wisconsin strain, Day 21 | 101 | 102 | 104 | 101
  B/Malaysia strain, Day 0 | 53 | 49 | 44 | 47
  B/Malaysia strain, Day 21 | 101 | 101 | 100 | 98
  B/Jiangsu strain, Day 0 | 33 | 40 | 45 | 41
  B/Jiangsu strain, Day 21 | 102 | 99 | 78 | 67

5. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of any specified solicited local symptoms reported irrespective of intensity grade. Grade 3 pain was defined as considerable pain that prevented normal activity. Grade 3 redness and swelling were defined as redness/swelling above 100 millimeters (mm).
Time Frame: During a 7 day (Days 0-6) follow-up period after vaccination
Population: Analysis was performed on theTotal Vaccinated cohort which included all subjects with a documented vaccine administration and symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 105 | 104 | 105 | 105
Subjects
  Any Pain | 76 | 79 | 74 | 52
  Grade 3 Pain | 0 | 2 | 3 | 0
  Any Redness | 3 | 6 | 5 | 1
  Grade 3 Redness | 0 | 0 | 0 | 0
  Any Swelling | 3 | 4 | 7 | 2
  Grade 3 Swelling | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms Reported by the Former GSK Rules of Grading.
Description: Solicited local symptoms assessed by the former GSK rules of grading were pain, redness and swelling. Any was defined as occurrence of any specified solicited local symptoms reported irrespective of intensity grade. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling were defined as redness/swelling above 50 millimeters (mm).
Time Frame: During a 7-day follow-up period (Days 0-6) after vaccination
Population: Analysis was performed on the Total Vaccinated cohort which included all subjects with a documented vaccine administration and symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 105 | 104 | 105 | 105
Subjects
  Any Pain | 76 | 79 | 74 | 52
  Grade 3 Pain | 0 | 2 | 3 | 0
  Any Redness | 3 | 6 | 5 | 1
  Grade 3 Redness | 1 | 2 | 1 | 0
  Any Swelling | 3 | 4 | 7 | 2
  Grade 3 Swelling | 1 | 2 | 3 | 1

7. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, headache, myalgia, nausea, shivering and fever. Any =occurrence of any specified solicited general symptoms reported irrespective of intensity grade or relationship to vaccination. Any fever = oral temperature ≥ 38.0 degrees Celsius (°C).. Grade 3 symptoms = symptoms that prevented normal activities. Grade 3 fever = oral temperature ≥39.0°C. Related = symptoms considered by the investigator to have a causal relationship to vaccination
Time Frame: During a 7-day follow-up period (Days 0-6) after vaccination
Population: as for outcome 5
Measure: Number; unit: Subjects
Groups:
- Trivalent Influenza Vaccine GSK 2115160A Group 2: Subjects in this group received 1full dose of GSK Biologicals' trivalent influenza vaccine, administered intramuscularly in the deltoid region of the non-dominant arm, at Day 0
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 105 | 104 | 105 | 105
Subjects
  Any Arthralgia | 6 | 25 | 13 | 12
  Grade 3 Arthralgia | 1 | 3 | 2 | 0
  Related Arthralgia | 6 | 25 | 13 | 11
  Any Fatigue | 33 | 47 | 36 | 34
  Grade 3 Fatigue | 2 | 4 | 3 | 1
  Related Fatigue | 32 | 47 | 36 | 33
  Any Headache | 25 | 36 | 28 | 26
  Grade 3 Headache | 3 | 2 | 1 | 1
  Related Headache | 24 | 33 | 26 | 23
  Any Myalgia | 17 | 40 | 33 | 15
  Grade 3 Myalgia | 1 | 3 | 3 | 1
  Related Myalgia | 17 | 40 | 33 | 15
  Any Nausea | 8 | 11 | 8 | 9
  Grade 3 Nausea | 2 | 2 | 2 | 1
  Related Nausea | 8 | 10 | 8 | 8
  Any Shivering | 4 | 10 | 9 | 4
  Grade 3 Shivering | 1 | 2 | 1 | 0
  Related Shivering | 4 | 10 | 9 | 4
  Any Fever | 1 | 3 | 2 | 1
  Grade 3 Fever | 0 | 0 | 0 | 0
  Related Fever | 1 | 3 | 2 | 1

8. Secondary Outcome: Number of Subjects With Any ,Grade 3 and Related Solicited General Symptoms Reported by the Former GSK Rules of Grading.
Description: Solicited general symptoms assessed by the former GSK rules of grading were arthralgia, fatigue, headache, myalgia, nausea, shivering and fever. Any = occurrence of any specified solicited general symptoms reported irrespective of intensity grade or relationship to vaccination. Any fever = oral temperature ≥ 37.5 °C. Grade 3 symptoms = symptoms that prevented normal activities. Grade 3 fever = oral temperature above 39.0°C. . Related = symptoms considered by the investigator to have a causal relationship to vaccination.
Time Frame: During a 7-day follow-up period (Days 0-6) after vaccination
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 105 | 104 | 105 | 105
Subjects
  Any Arthralgia | 6 | 25 | 13 | 12
  Grade 3 Arthralgia | 1 | 3 | 2 | 0
  Related Arthralgia | 6 | 25 | 13 | 11
  Any Fatigue | 33 | 47 | 36 | 34
  Grade 3 Fatigue | 2 | 4 | 3 | 1
  Related Fatigue | 32 | 47 | 36 | 33
  Any Headache | 25 | 36 | 28 | 26
  Grade 3 Headache | 3 | 2 | 1 | 1
  Related Headache | 24 | 33 | 26 | 23
  Any Myalgia | 17 | 40 | 33 | 15
  Grade 3 Myalgia | 1 | 3 | 3 | 1
  Related Myalgia | 17 | 40 | 33 | 15
  Any Nausea | 8 | 11 | 8 | 9
  Grade 3 Nausea | 2 | 2 | 2 | 1
  Related Nausea | 8 | 10 | 8 | 8
  Any Shivering | 4 | 10 | 9 | 4
  Grade 3 Shivering | 1 | 2 | 1 | 0
  Related Shivering | 4 | 10 | 9 | 4
  Any Fever | 1 | 2 | 2 | 1
  Grade 3 Fever | 0 | 0 | 0 | 0
  Related Fever | 1 | 2 | 2 | 1

9. Secondary Outcome: Number of Subjects Reporting Any Medically Significant Conditions (MSCs) and Auto-immune Diseases (AIDs).
Description: MSCs were defined as those adverse events (AEs) prompting emergency room visits, hospitalizations or physician visits and that were not routine visits for physical examination or vaccination. AIDs include a large group of diseases characterized by abnormal functioning of the immune system that causes immune system to produce antibodies against own tissues.
Time Frame: During the entire study period (Days 0-180)
Population: Analysis was performed on the Total Vaccinated cohort which included all subjects with a documented vaccine administration.
Measure: Number; unit: Subjects
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 105 | 105 | 105 | 105
Subjects
  MAE(s) | 1 | 4 | 5 | 5
  AID | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AE(s).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination
Time Frame: During a 21 day (Days 0-20) follow-up period after vaccination-
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 105 | 105 | 105 | 105
Subjects
  Any unsolicited AE(s) | 7 | 7 | 16 | 11
  Grade 3 unsolicited AE(s) | 0 | 1 | 3 | 2
  Related unsolicited AE(s) | 3 | 3 | 7 | 3

11. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Days 0-180)
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Number analyzed (Participants) | 105 | 105 | 105 | 105
Subjects
  Any SAE(s) | 0 | 0 | 0 | 1.0
  Related SAE(s) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): During the entire study period i.e. Day 0 to Day 180 ; Solicited local and general symptoms: During Day 0- Day 6 post vaccination period.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 | Trivalent Influenza Vaccine GSK 2115160A Group 1 | Trivalent Influenza Vaccine GSK 2115160A Group 2
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/105 | 0/105 | 1/105
Other Adverse Events (participants affected / at risk) | 84/105 | 90/105 | 81/105 | 72/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 (N=105) | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 (N=105) | Trivalent Influenza Vaccine GSK 2115160A Group 1 (N=105) | Trivalent Influenza Vaccine GSK 2115160A Group 2 (N=105)
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quadrivalent Influenza Vaccine GSK 2115160A Group 1 (N=105) | Quadrivalent Influenza Vaccine GSK 2115160A Group 2 (N=105) | Trivalent Influenza Vaccine GSK 2115160A Group 1 (N=105) | Trivalent Influenza Vaccine GSK 2115160A Group 2 (N=105)
Pain (General disorders) | 76 | 79 | 74 | 52
Redness (General disorders) | 3 | 6 | 5 | 1
Swellling (General disorders) | 3 | 4 | 7 | 2
Arthralgia (General disorders) | 6 | 25 | 13 | 12
Fatigue (General disorders) | 33 | 47 | 36 | 34
Headache (General disorders) | 25 | 36 | 28 | 26
Myalgia (General disorders) | 17 | 40 | 33 | 15
Nausea (General disorders) | 8 | 11 | 8 | 9
Shivering (General disorders) | 4 | 10 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.